CLINICAL TRIAL: NCT06029270
Title: A Randomized Phase II Study of Nivolumab Versus Nivolumab and BMS-986016 (Relatlimab) as Maintenance Treatment After First-Line Treatment With Platinum-Gemcitabine-Nivolumab for Patients With Epstein-Barr Virus-Associated Recurrent/Metastatic Nasopharyngeal Carcinoma (REMAIN)
Brief Title: Testing the Addition of BMS-986016 (Relatlimab) to the Usual Immunotherapy After Initial Treatment for Recurrent or Metastatic Nasopharyngeal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-06678; NCI-2023-06678 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN011 (Other: NRG Oncology); NRG-HN011 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2023-09-07; First posted 2023-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Nasopharyngeal Carcinoma; Recurrent Nasopharyngeal Carcinoma; Stage IV Nasopharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Magnetic Resonance Spectroscopy; Nivolumab; relatlimab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (Nivolumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes. Cycles repeat every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI on study. Patients also undergo PET/CT or bone scan as clinically indicated.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography
- Arm II (Nivolumab, relatlimab) (Experimental): Patients receive nivolumab IV over 30 minutes and relatlimab IV over 30-90 minutes. Cycles repeat every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI on study. Patients also undergo PET/CT or bone scan as clinically indicated.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Biological: Relatlimab
- Induction therapy (Platinum-gemcitabine-nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 of each cycle, cisplatin IV or carboplatin IV over 30-60 minutes on day 1 of each cycle and gemcitabine IV over 30 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI and blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Induction therapy (Platinum-gemcitabine-nivolumab)
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
  Arms: Arm I (Nivolumab); Arm II (Nivolumab, relatlimab)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Induction therapy (Platinum-gemcitabine-nivolumab)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Induction therapy (Platinum-gemcitabine-nivolumab)
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Induction therapy (Platinum-gemcitabine-nivolumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: Arm I (Nivolumab); Arm II (Nivolumab, relatlimab)
Biological: Relatlimab — Given IV
  Other Names: BMS 986016; BMS-986016; BMS986016; Immunoglobulin G4, Anti-(human Lymphocyte Activation Gene-3 Protein) (Human Heavy Chain), Disulfide with Human Light Chain, Dimer
  Arms: Arm II (Nivolumab, relatlimab)

SUMMARY:
This phase II trial tests the addition of BMS-986016 (relatlimab) to the usual immunotherapy after initial treatment for nasopharyngeal cancer that has come back after a period of improvement (recurrent) or that has spread from where it first started (primary site) to other places in the body (metastatic). Relatlimab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. The usual approach of treatment is initial treatment with chemotherapy such as the combination of cisplatin (or carboplatin) and gemcitabine, along with immunotherapy such as nivolumab. After the initial treatment is finished, patients may continue to receive additional immunotherapy. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Gemcitabine is a chemotherapy drug that blocks the cells from making deoxyribonucleic acid (DNA) and may kill cancer cells. Giving BMS-986016 in addition to the usual immunotherapy after initial treatment may extend the time without the tumor cells growing or spreading longer than the usual approach in patients with recurrent or metastatic nasopharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if adding BMS-986016 (relatlimab) to nivolumab maintenance therapy shows a signal of improved progression-free survival (PFS) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in patients who do not progress following treatment with platinum-gemcitabine-nivolumab combination in the first-line treatment of recurrent and/or metastatic nasopharyngeal carcinoma (R/M NPC).

SECONDARY OBJECTIVES:

I. To determine if adding BMS-986016 (relatlimab) to nivolumab maintenance improves overall survival (OS) compared to nivolumab maintenance alone.

II. To compare patterns of failure (local-regional relapse and distant metastasis) between treatment arms.

III. To determine if adding BMS-986016 (relatlimab) to nivolumab maintenance improves objective response, duration of response, and disease control rate compared to nivolumab maintenance alone.

IV. To evaluate the tolerability of nivolumab-BMS-986016 (relatlimab) maintenance and assess and compare toxicity between arms based on the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) criteria.

V. To evaluate baseline plasma Epstein-Barr virus (EBV) DNA (< 2000 copies/mL versus [vs.] >= 2000 copies/mL) as a prognostic biomarker.

VI. To validate post-induction plasma EBV DNA (detectable [>= 1 copies/mL] vs. undetectable [0 copies/mL]) as a prognostic biomarker.

EXPLORATORY OBJECTIVES:

I. To collect blood and tissue specimens for future translational science studies.

II. To assess post-induction plasma EBV DNA (detectable [>= 1 copies/mL] vs. undetectable [0 copies/mL]) as a predictive biomarker.

OUTLINE:

INDUCTION THERAPY: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 of each cycle, cisplatin IV or carboplatin IV over 30-60 minutes on day 1 of each cycle and gemcitabine IV over 30 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood sample collection during screening and on study.

MAINTENANCE THERAPY: Patients who do not progress radiologically are randomized to 1 of 2 arms.

ARM I: Patients receive nivolumab IV over 30 minutes. Cycles repeat every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI on study. Patients also undergo positron emission tomography (PET)/CT or bone scan as clinically indicated.

ARM II: Patients receive nivolumab IV over 30 minutes and relatlimab IV over 30-90 minutes. Cycles repeat every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI on study. Patients also undergo PET/CT or bone scan as clinically indicated.

After completion of study treatment, patients are followed up every 4 months for 2 years, every 6 months in years 3-5, and then annually.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION:
* Pathologically (histologically or cytologically) proven diagnosis of nasopharyngeal carcinoma (NPC) that has recurred locoregionally and/or is present at distant sites. Patients who present with metastatic disease (de novo) at diagnosis are also eligible. For locoregional recurrence, the disease must not be amenable to potentially curative surgery or re-irradiation. Eligible patient must have the following characteristics:

  * Tumor showing (histological/cytological) Epstein-Barr encoded ribonucleic acid (EBER)-positivity (e.g., In situ hybridization, immunohistochemistry) or
  * A known history of detectable plasma EBV DNA (via a polymerase chain reaction [PCR]-based assay) at any time point since the initial diagnosis of NPC.
* Measurable disease as defined by RECIST 1.1 criteria. Lesion(s) that have been irradiated previously can be counted as measurable as long as radiological progression after the prior radiation therapy has been demonstrated.

  * Contrast enhanced CT scan of the chest. The contrast enhanced CT component of a whole-body PET-CT is also acceptable. The plain (non-contrast) CT component of a PET-CT is not acceptable.
  * CT the abdomen and pelvis, if clinically indicated (diagnostic quality with contrast, unless contraindicated).
  * Patients with known locoregional disease must have contrast enhanced MRI or CT of the nasopharynx and neck as this disease site(s) may be assessed as target lesions. For patients without known locoregional disease, imaging of the nasopharynx and neck is optional.
  * Symptomatic and active brain metastases and/or leptomeningeal metastasis on CT and/or MRI imaging: Patients who have prior therapies for brain and leptomeningeal metastasis or cord/cauda compression who are clinically stable for >= 2 months prior to registration and have discontinued systemic steroids therapy (> 10 mg/day prednisone or equivalent) > 4 weeks prior to registration are eligible.
  * Patients with base of skull involvement by NPC are allowed unless their disease is directly invading the brain parenchyma, associated with clinical symptoms and/or significant vasogenic edema on radiological imaging.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status of 0-2.
* Negative urine or serum pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal.
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3.
* Platelets >= 100,000 cells/mm^3.
* Hemoglobin (Hgb) >= 8.0 g/dL (Transfusion is accepted. Erythropoietin dependency not accepted.).
* Total bilirubin =< 1.5 × institutional upper limit of normal (ULN) or direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 × ULN. Patients with known Gilbert's disease who have serum bilirubin level =< 3 × ULN may be enrolled.
* Alanine transaminase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 × ULN (=< 5 × ULN for patients with liver metastases).
* Serum creatinine =< 1.5 × ULN or calculated creatinine clearance (CrCl) based on Cockcroft-Gault equation >= 30 mL/min for patients with serum creatinine levels > 1.5 × ULN. Cisplatin or carboplatin may be used at the discretion of the investigator - except for patients with CrCl between 30-50 mL/min, for whom carboplatin should be used instead of cisplatin. CrCl must be > 50 mL/min for cisplatin to be used.
* Albumin-adjusted calcium level based on corrected calcium equation =< 1.5 × ULN (patients are allowed to have treatment for hypercalcemia prior to starting treatment).
* No prior systemic treatment for recurrent/metastatic (R/M) NPC including cytotoxic chemotherapy. Prior treatment for non-recurrent and non-metastatic NPC is allowed.
* No prior treatment with a PD-1 inhibitor (except if given as adjuvant or neoadjuvant therapy for NPC), PD-L1 inhibitor, anti-PD-L2 inhibitor, LAG-3 inhibitor, CTLA-4 inhibitor (except if given as adjuvant or neoadjuvant therapy for non-recurrent and non-metastatic NPC), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* The interval between the last dose of curative-intent treatment for non-recurrent, non-metastatic NPC, including definitive radiotherapy (RT) and/or induction, concurrent, or adjuvant chemotherapy and recurrence must be ˃ 6 months.
* Clinically significant toxicities from any prior systemic therapy or radiotherapy must have resolved to grade 0 or 1 as per National Cancer Institute (NCI) CTCAE v 5.0 - except alopecia, dry mouth, dysgeusia, dysphagia, and fatigue. Patients with a history of grade 3-4 cisplatin related neuropathy must have recovered to grade 0-2 prior to registration. Patients with a history of hearing impairment, or ototoxicity from prior cisplatin, of any grade are allowed.
* No prior palliative RT within 30 days prior to registration. This includes RT given with palliative intent to recurrent/metastatic sites. The irradiated sites must not be the only sites of measurable recurrent disease.
* No major surgical procedures within 30 days prior to registration.
* No history of unstable angina requiring hospitalization within the last 6 months.
* No history of myocardial infarction within the last 6 months.
* New York Heart Association Functional Classification II or better (New York Heart Association [NYHA] Functional Classification III/IV are not eligible). Patients with symptomatic coronary artery disease, congestive heart failure or a known history of having a left ventricular ejection fraction < 50% must be stably controlled with medication in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* No prior history of myocarditis.
* No active infection requiring IV antibiotics, IV antiviral, or IV antifungal treatments at the time of study registration.
* No history of (non-infectious) pneumonitis that required steroids or current pneumonitis requiring steroids and/or immunosuppressive therapy, idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans), or idiopathic pneumonitis.
* No history of multi-drug resistant mycobacterium tuberculosis (TB) or active TB, as defined by systemic treatment received =< 2 years prior to registration. Note: Patients who had a history of treated TB ˃ 2 years prior to registration are allowed.
* No prior solid organ transplant or bone marrow transplant.
* No conditions requiring systemic treatment with either immunosuppressive doses of corticosteroids (> 10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days of registration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Steroid premedication for the prophylaxis of CT contrast-related allergies is allowed. The use of dexamethasone as an anti-emetic premedication prior to chemotherapy is also allowed.
* No active autoimmune disease requiring systemic treatment (i.e., disease modifying agents, corticosteroids, or immunosuppressive drugs) within the past 2 years. These may include (but not limited to) patients with a history of immune-related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), rheumatoid arthritis, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's disease, ulcerative colitis, autoimmune hepatitis, glomerulonephritis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome.

  * Note: Patients are permitted to enroll if they have vitiligo; type I diabetes mellitus; hypothyroidism, pituitary or adrenal insufficiency requiring only hormone replacement; alopecia; and/or psoriasis not requiring systemic treatment. Conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* No prior live vaccine within 30 days prior to registration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist [registered trademark]) are live attenuated vaccines and are not allowed. Coronavirus disease 2019 (COVID-19) vaccines that are approved by the local drug regulatory authority of the participating region are allowed.
* No known history of grade 3-4 allergic reaction or hypersensitivity reaction to cisplatin, carboplatin, or gemcitabine.
* No known history of grade 4 hypersensitivity (or infusion) reaction to any monoclonal antibody. Patients who had prior grade 3 hypersensitivity (or infusion) reaction but could tolerate resumption of the antibody treatment after appropriate pre-medication are eligible.
* PRIOR TO STEP 2 REGISTRATION:
* Collection of plasma EBV DNA at baseline is mandatory for all patients prior to Step 2 registration and induction treatment.

  * Note: Submission of the baseline sample will be batch shipped.
* PRIOR TO STEP 3 REGISTRATION/RANDOMIZATION: PATIENTS WITHOUT PROGRESSIVE DISEASE (PD) ONLY:
* All patients must have received minimum of 3 cycles, and up to a maximum of 6 cycles of induction treatment within 20 weeks from cycle 1, day 1 of induction treatment (i.e., patients must have completed all induction treatment within 20 weeks from cycle 1 day 1, including the treatment breaks). Patients must have completed 6 cycles of induction treatment, except in the following circumstances:

  * Significant dose delays as a result of treatment-related toxicities.
  * Intercurrent illness(s), that rendered the patient unable to continue induction treatment.
  * Note: If a patient received < 6 cycles of induction treatment for reasons other than the above circumstances, they will not be eligible for randomization.
* A CT scan within 30 days prior to Step 3 registration/randomization is required. If the most recent scan performed is not within this time frame, a repeat scan is required to assess response.
* Did not meet any criteria that result in permanent discontinuation of study treatment during induction treatment phase.
* Must meet the criteria for starting/resuming a new cycle of maintenance treatment.
* Did not experience any nivolumab-related autoimmune toxicities that would result in permanent discontinuation of nivolumab during the induction treatment phase.
* Collection of the plasma EBV DNA post-induction treatment is mandatory.

  * Note: Submission of the post-induction sample will be batch shipped.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from randomization to progressive disease (PD) or death due to any cause, assessed up to 6 years
  Will be assessed in both treatment arms and will be estimated using the Kaplan-Meier method. The comparison of PFS distributions between treatment arms will be performed using the log-rank test. Additional analyses of treatment effect will be performed using Cox models with the stratification factors included as a fixed covariates, as well as other tumor and patient characteristics, listed below. Median PFS and the corresponding 95% confidence intervals (CIs) for each arm will be estimated with the Brookmeyer-Crowley method. Multivariable analysis will be performed using a Cox proportional hazards model and relevant patient and tumor characteristics (country [Asian sites versus (vs.) Non-Asian sites], keratinizing squamous carcinoma, sex, age, and baseline Epstein-Barr virus (EBV) deoxyribonucleic acid [DNA]). Hazard ratios and their respective 85% lower confidence bound, and 95% confidence intervals will be provided.

SECONDARY OUTCOMES:
Overall survival (OS) | Time from randomization to death due to any cause, assessed up to 6 years
  Will be estimated using the Kaplan-Meier method and between-arm differences will be assessed using the log-rank test. Median OS and the corresponding 95% CIs using log-log transformation to survival function for each arm will be estimated with the Brookmeyer-Crowley method.
Tumor response | Up to 6 years
  Will be assessed using Response Evaluation Criteria in Solid Tumors version 1.1. Cox proportional hazards models will be used to determine hazard ratios (cause-specific hazard ratios in the case of endpoints with competing risks) and to assess the effects of covariates of interest. Fine-Gray sub-distribution hazards Cox model will be used to complement the competing risk analyses.
Locoregional failure | Up to 6 years
  Cox proportional hazards models will be used to determine hazard ratios (cause-specific hazard ratios in the case of endpoints with competing risks) and to assess the effects of covariates of interest. Fine-Gray sub-distribution hazards Cox model will be used to complement the competing risk analyses.
Distant metastasis | Up to 6 years
  Cox proportional hazards models will be used to determine hazard ratios (cause-specific hazard ratios in the case of endpoints with competing risks) and to assess the effects of covariates of interest. Fine-Gray sub-distribution hazards Cox model will be used to complement the competing risk analyses.
Incidence of adverse events (AEs) | Up to 6 years
  Will be graded using Common Terminology Criteria for Adverse Events version 5.0. Counts of all AEs by grade will be provided by treatment arm. Counts and frequencies will be provided for the worst grade AE experienced by the patient by treatment arm. The rate of patients with at least 1 grade 3 or higher AE will be compared between the treatment arms using a chi-square test for proportions and confidence intervals for rate difference will be computed using Miettinen-Nurminen (score) method
Post-induction plasma EBV DNA as a prognostic biomarker | Up to 6 years
  Will be defined as a binary biomarker (detectable: >= 1 copies/mL vs. undetectable: 0 copies/mL). Biomarker effect HRs from multivariable Cox models, including key tumor and patient characteristics will also be reported.
Pre-induction plasma EBV DNA vs. progressive disease (PD) during induction treatment | Up to 6 years
  Will include all patients treated with concurrent (induction) treatment and a binary biomarker based on pre-induction plasma EBV DNA (< 2000 vs. ≥2000 copies/mL). PD rates during induction for each biomarker subgroup will be computed assuming a binomial distribution and compared between biomarker subgroups using a chi-square test. Multivariable Cox models, including key tumor and patient characteristics will also be included.
Persistent plasma EBV DNA vs. PFS | Up to 6 years
  Will examine the association between persistent EBV DNA after induction treatment and PFS. Only randomized patients with positive pre-induction plasma EBV DNA will be included (~90-95%). Patients will be classified into "EBV DNA positive to negative" and "EBV DNA consistently positive" based on the pre-induction and post-induction EBV DNA. Multivariable Cox models, including key tumor and patient characteristics will also be included.

OTHER OUTCOMES:
Post-induction EBV DNA as a predictive biomarker | Up to 6 years
  Will be assessed of the predictive role of post-induction EBV DNA on PFS and OS will be performed using the binary biomarker. Cox proportional hazards model with treatment arm, binary biomarker, and its interaction will be used for these analyses. Treatment effect hazard ratios and 95% confidence intervals will be reported. Adjusted HR estimates will be obtained after adding key patient and tumor characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Brigette B Ma, Principal Investigator — NRG Oncology
Locations (77):
- United States (72):
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MEJ, Council Bluffs, Iowa
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm